CLINICAL TRIAL: NCT06802809
Title: Evaluation of the Efficacy of Lactobacillus Crispatus M247 Administration in Promoting Clearance of Genital HR-HPV Infection and Modulating the Vaginal Microbiota: A Multicenter, Randomized, Placebo-Controlled, Single-Blind, Longitudinal, Prospective Clinical Trial
Brief Title: Efficacy of Probiotic Lactobacillus Crispatus M247 in Promoting High-risk Human Papillomavirus (HR-HPV) Infection Clearance and Modifying Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol n° 774/18.10.2021/AK
Record Dates: First submitted 2025-01-25; First posted 2025-01-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Experimental, multicenter, randomized, placebo-cntrolled, longitudinal, prospective, single-blind, parallel-group study.
Who Masked: Participant
Masking Description: Single-blind design (participants unaware of their group allocation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement Lactobacillus crispatus M247 group (Experimental): Participants in this group will receive probiotic supplement Lactobacillus crispatus M247 (Crispact®) in stick form, administered orally at a dose of one stick per day for 4 months. Each stick contains 20 billion CFU of L. crispatus M247.
  Interventions: Dietary Supplement: Lactobacillus crispatus M247 (Crispact®)
- Control Group (Placebo Comparator): Participants in the control group will receive a placebo identical in appearance and packaging to the experimental product, administered orally at a dose of one stick per day for 4 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus crispatus M247 (Crispact®) — Crispact® is a probiotic food supplement containing Lactobacillus crispatus M247.
  Arms: Probiotic supplement Lactobacillus crispatus M247 group
Other: Placebo — The placebo does not contain the active probiotic strain and consists of inactive excipients.
  Arms: Control Group

SUMMARY:
This clinical trial evaluates the efficacy of the probiotic strain Lactobacillus crispatus M247 in promoting the clearance of genital high-risk human papillomavirus (HR-HPV) infection and restoring the balance of the vaginal microbiota. The study adopts a multicenter, randomized, single-blind, longitudinal, prospective design involving HR-HPV-positive patients. Primary outcomes include HR-HPV clearance rates and microbiota composition changes.

DETAILED DESCRIPTION:
This study investigates the potential benefits of Lactobacillus crispatus M247, a probiotic strain with proven ability to promote vaginal health, in the management of HR-HPV infections. Lactobacillus crispatus M247 has demonstrated superior probiotic properties, including the ability to produce lactic acid and hydrogen peroxide, which contribute to maintaining a stable vaginal microbiota and potentially inhibiting HR-HPV persistence.

Participants will be randomized to receive either Lactobacillus crispatus M247 or a placebo over a specified study period. The primary aim is to evaluate the probiotic's efficacy in enhancing HR-HPV clearance rates and restoring a balanced vaginal microbiota. Secondary objectives include assessing changes in cervical cytology and participant-reported outcomes on vaginal health. By focusing exclusively on the role of Lactobacillus crispatus M247, the study seeks to establish its clinical relevance in HR-HPV management and its potential as a therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-69 years.
* First diagnosis of HR-HPV infection via DNA-HPV screening.
* Cytology results showing ASC-US or LSIL.
* Negative colposcopy or biopsy (absence of lesions).
* Ability to provide written informed consent.

Exclusion Criteria:

* Prior HPV vaccination.
* History of cervical treatments for pre-neoplastic pathology.
* Cytology showing HSIL (High-Grade Squamous Intraepithelial Lesion) requiring treatment.
* Current treatment with antibiotics, immunomodulatory, or immunosuppressive therapies.
* Diagnosed immune system or neoplastic diseases requiring chemotherapy.
* Pregnancy, lactation, or planning to become pregnant within 6 months.
* Known hypersensitivity to product components.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes individuals who self-identify as female and meet the inclusion criteria, as the study focuses on conditions affecting the female reproductive system (e.g., HR-HPV infections and vaginal microbiota.
Enrollment: 66 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
HR-HPV Clearance Rate | Baseline to 4 months post-intervention
  Percentage of participants in whom HR-HPV infection is no longer detectable, as assessed by an HPV-DNA test.

SECONDARY OUTCOMES:
Modifications in Vaginal Microbiota | Baseline to 4 months post-intervention.
  Changes in the composition of the vaginal microbiota, including the abundance of Lactobacillus species (especially Lactobacillus crispatus) and microbiota diversity indices, as assessed by Next-Generation Sequencing of the 16S ribosomal RNA gene (NGS 16S) sequencing.
Microbiota Characteristics Favoring HR-HPV Infection or Clearance | Baseline to 4 months post-intervention.
  Identification of vaginal microbiota profiles (e.g., CST-I (Community State Type-I) to CST-IV (Community State Type-IV) distribution) associated with HR-HPV persistence or clearance, as determined by NGS 16S sequencing
Cervical Cytology Normalization | Baseline to 4 months post-intervention.
  Proportion of participants with normalization of cervical cytology results, transitioning from ASC-US (Atypical Squamous Cells of Undetermined Significance) or LSIL (Low-Grade Squamous Intraepithelial Lesion) to normal cytology, as determined by Papanicolaou (Pap) test analysis.
Number of patients reporting side effects to probiotic Crispact® intake | From baseline to 4 months post-intervention.
  Number and type of adverse events reported, including gastrointestinal symptoms, allergic reactions, or other health concerns, as recorded in participant safety logs.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico-San Marco", Catania
  - Nuovo Ospedale di Lentini, Lentini
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone" di Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No